CLINICAL TRIAL: NCT04328441
Title: Reducing Health Care Workers Absenteeism in COVID-19 Pandemic by Enhanced Trained Immune Responses Through Bacillus Calmette-Guérin Vaccination, a Randomized Controlled Trial.
Brief Title: Reducing Health Care Workers Absenteeism in Covid-19 Pandemic Through BCG Vaccine
Acronym: BCG-CORONA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, MJM Bonten, Prof. M.J.M. Bonten, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL73249.041.20
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: COVID-19
Keywords: Health care workers
MeSH Terms: conditions — COVID-19 | interventions — BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinded are the pharmacist and the research nurse that administers the study medication. These persons are not involved in the further conduction of the trial or in the assessment of outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BCG vaccine (Experimental): Intracutaneously 0.1ml BCG vaccine, which accounts for 0.075mg of attenuated Mycobacterium bovis.
  Interventions: Drug: BCG Vaccine
- Placebo (Placebo Comparator): Intracutaneously 0.1ml of 0.9% NaCl solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BCG Vaccine — Intracutaneously 0.1ml BCG vaccine, which accounts for 0.075mg of attenuated Mycobacterium bovis
  Other Names: Danish strain 1331
  Arms: BCG vaccine
Drug: Placebo — Intracutaneously 0.1ml NaCl 0,9%
  Other Names: NaCl 0,9%
  Arms: Placebo

SUMMARY:
Rationale: Covid-19 spreads rapidly throughout the world. A large epidemic in the Netherlands would seriously challenge the available hospital capacity, and this would be augmented by absenteeism of healthcare workers (HCW). Strategies to prevent absenteeism of HCW are, therefore, desperately needed to safeguard continuous patient care. Bacille Calmette-Guérin (BCG) is a vaccine against tuberculosis, with protective non-specific effects against other respiratory tract infections in in vitro and in vivo studies, and reported significant reductions in morbidity and mortality. The hypothesis is that BCG vaccination can reduce HCW absenteeism during the epidemic phase of Covid-19.

Objective: Primary objective: To reduce absenteeism among HCW with direct patient contacts during the epidemic phase of Covid-19. Secondary objective: To reduce hospital admission, ICU admission or death in HCW with direct patient contacts during the epidemic phase of Covid-19.

Study design: A placebo-controlled adaptive multi-centre randomized controlled trial.

Study population: HCW with direct patient contacts among which nurses and physicians working at emergency rooms and wards where Covid-19-infected patients are treated.

Intervention: Participants will be randomized between intracutaneous administration of BCG vaccine or placebo in a 1:1 ratio.

Main study parameters/endpoints: Primary endpoint: number of days of (unplanned) absenteeism for any reason. Secondary endpoints include the number of days of (unplanned) absenteeism because of documented Covid-19 infection, and the cumulative incidence of hospital admission, Intensive Care Admission, and death.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Based on previous experience and randomized controlled trials in adult and elderly individuals, the risks of BCG vaccination are considered low. The objective of this trial is to evaluate the beneficial effects of BCG vaccination through a lower work absenteeism rate of HCW and/or a mitigated clinical course of Covid-19 infection. The primary endpoint and the adaptive design with frequent interim analyses facilitate maximum efficiency of the trial, so that results can inform policy making during the ongoing epidemic.

DETAILED DESCRIPTION:
Since the beginning of 2020, SARS-CoV-2 spread rapidly throughout China and the rest of the world, with on 27 February 2020 the first detected case in the Netherlands.

According to the WHO, Health-care workers (HCW) face an elevated risk of exposure to - and infection of Covid-19.

Bacillus Calmette-Guérin (BCG) was developed as a vaccine against tuberculosis, but studies have shown its ability to induce potent protection against other infectious diseases: the so called non-specific effects (NSEs). A favorable in vitro or in vivo effect has been observed in studies for distinct viral pathogens, e.g. respiratory syncytial virus, yellow fever, herpes simplex virus; human papilloma virus.

Based on the capacity of BCG to reduce the incidence of respiratory tract infections in children, to exert antiviral effects in experimental models; and to reduce viremia in an experimental human model of viral infection, the hypothesis is that BCG vaccination induces (partial) protection against susceptibility to and/or severity of Covid-19 infection. This study evaluates the efficacy of BCG to improve the clinical course of Covid-19 infection and to prevent absenteeism in order to safeguard continuous patient care.

This randomized controlled trial has been designed as a pragmatic study with a highly feasible primary endpoint, which is unplanned absenteeism, that can be continuously measured on a bi-weekly basis). This allows for the most rapid identification of a beneficial outcome that would allow other HCWs to also benefit from the intervention if and as soon as it has been demonstrated to be effective.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Male or female
* Hospital personnel (expected to) taking care for patients with SARS CoV-2 infection

Exclusion Criteria:

* Known allergy to (components of) the BCG vaccine or serious adverse events to prior BCG administration
* Known active or latent Mycobacterium tuberculosis or with another mycobacterial species. A history with- or a suspicion of M. tuberculosis infection.
* Fever (>38 C) within the past 24 hours
* Pregnancy
* Suspicion of active viral or bacterial infection
* Vaccination in the past 4 weeks or expected vaccination during the study period, independent of the type of vaccination.
* Severely immunocompromised subjects. This exclusion category comprises: a) subjects with known infection by the human immunodeficiency virus (HIV-1); b) neutropenic subjects with less than 500 neutrophils/mm3; c) subjects with solid organ transplantation; d) subjects with bone marrow transplantation; e) subjects under chemotherapy; f) subjects with primary immunodeficiency; g) severe lymphopenia with less than 400 lymphocytes/mm3; h) treatment with any anti-cytokine therapies. i) treatment with oral or intravenous steroids defined as daily doses of 10mg prednisone or equivalent for longer than 3 months, or probable use of oral or intravenous steroids in the following four weeks
* Active solid or non-solid malignancy or lymphoma within the prior two years
* Direct involvement in the design or the execution of the BCG-CORONA study
* Expected absence from work of ≥4 of the following 12 weeks due to any reason (holidays, maternity leave, retirement, planned surgery etc)
* Employed to the hospital < 22 hours per week
* Not in possession of a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1511 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Health Care Workers absenteeism | Maximum of 365 days
  Number of days of unplanned absenteeism for any reason

SECONDARY OUTCOMES:
the cumulative incidence of documented COVID-19 | Maximum of 365 days
the cumulative incidence of Hospital Admission due to documented COVID-19 | Maximum of 365 days
the number of days of unplanned absenteeism, because of documented COVID-19 | Maximum of 365 days
the cumulative incidence of self-reported acute respiratory symptoms or fever | Maximum of 365 days
the cumulative incidence of death due to documented COVID-19 | Maximum of 365 days
the cumulative incidence of Intensive Care Admission due to documented COVID-19 | Maximum of 365 days
the number of days of absenteeism, because of imposed quarantine as a result of exposure to COVID-19 | Maximum of 365 days
  Exploratory
the number of days of absenteeism, because of imposed quarantine as a result of having acute respiratory symptoms, fever or documented COVID-19 | Maximum of 365 days
  Exploratory
the number of days of unplanned absenteeism because of self-reported acute respiratory symptoms | Maximum of 365 days
  Exploratory
the number of days of self-reported fever (≥38 gr C) | Maximum of 365 days
  Exploratory
the cumulative incidence of self-reported fever (≥38 gr C) | Maximum of 365 days
  Exploratory
the number of days of self-reported acute respiratory symptoms | Maximum of 365 days
  Exploratory
the cumulative incidence of self-reported acute respiratory symptoms | Maximum of 365 days
  Exploratory
the cumulative incidence of death for any reason | Maximum of 365 days
  Exploratory
the cumulative incidence of Intensive Care Admission for any reason | Maximum of 365 days
  Exploratory
the cumulative incidence of Hospital Admission for any reason | Maximum of 365 days
  Exploratory
the cumulative incidence and magnitude of plasma/serum antibodies (IgA,M,G) and SARS-CoV-2-specific antibodies at 12 weeks after vaccination and at the end of the study period | Maximum of 365 days
  Exploratory
the cumulative incidence and magnitude of plasma/serum antibodies (IgA,M,G) and SARS-CoV-2-specific antibodies at 12 weeks after vaccination and at the end of the study period | 3-6 months after inclusion
  Exploratory

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bonten, MD, PhD, Principal Investigator — UMC Utrecht
Locations (9):
- Netherlands (9):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Radboud UMC, Nijmegen, Gelderland
  - Sint Maartenskliniek, Nijmegen, Gelderland
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch, North Brabant
  - Noordwest Ziekenhuisgroep locatie Alkmaar, Alkmaar, North Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Erasmus Medical Center, Rotterdam, South Holland
  - Hagaziekenhuis, The Hague, South Holland
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
The results of this study will be disclosed unreservedly at the end of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The content of the study protocol is published. The statistical analysis plan is attached. The informed consent form (in Dutch) could be obtained by sending a mail to one of the contact persons.
  The clinical study report and analytic code could be obtained by sending a mail to one of the contact persons after publication of the study in a peer-reviewed journal.

REFERENCES:
- [Derived] Ten Doesschate T, Moorlag SJCFM, van der Vaart TW, Taks E, Debisarun P, Ten Oever J, Bleeker-Rovers CP, Verhagen PB, Lalmohamed A, Ter Heine R, van Crevel R, van de Wijgert J, Janssen AB, Bonten MJ, van Werkhoven CH, Netea MG; BCG-CORONA study team#. Two Randomized Controlled Trials of Bacillus Calmette-Guerin Vaccination to reduce absenteeism among health care workers and hospital admission by elderly persons during the COVID-19 pandemic: A structured summary of the study protocols for two randomised controlled trials. Trials. 2020 Jun 5;21(1):481. doi: 10.1186/s13063-020-04389-w. PMID 32503602

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-05-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT04328441/SAP_000.pdf